CLINICAL TRIAL: NCT02214485
Title: Integrated Care and Lower Extremity Strength Training Among Community-Dwelling Frail Older Adults in Taiwan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 201101038RC
Record Dates: First submitted 2013-09-30; First posted 2014-08-12 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Frailty
Keywords: frailty; exercise; intervention
MeSH Terms: conditions — Frailty; Motor Activity | interventions — Delivery of Health Care, Integrated

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- integrated care (IC) (Experimental): Subjects will receive such care twice weekly for 12 weeks.
  Interventions: Behavioral: integrated care
- lower extremity strength training (LEST) (Experimental): Subjects will receive training twice weekly for 12 weeks
  Interventions: Behavioral: lower extremity strength training

INTERVENTIONS:
Behavioral: integrated care — Participants visit the study site with health education, social activities, warm up, stretch, and low intensity resistance exercise for about 1 hour per week. If any medical problems or functional decline suspected during the visit, the case manager refers participants to their primary care physicians for further managements.
  Arms: integrated care (IC)
Behavioral: lower extremity strength training — Participants receive 2 sessions of 30-minute lower extremity strength straining using isotonic strength training machines each week. The intensity is set at 60-80% of 1 repetition maximum (RM). Evaluation of the exercise protocol are repeated every 2 weeks for individualized adjustments.
  Arms: lower extremity strength training (LEST)

SUMMARY:
Objective: To determine the differential effectiveness of integrated care (IC) and lower extremity strength training (LEST) among community-dwelling frail older adults in Taiwan.

Method: The investigators randomize participants at Bei-Hu site from the "Intervention study of Geriatric Frailty, Osteoporosis, and Depression in a Community Based Randomized Trial" into 12 weeks of either IC or LEST. Outcome assessments are performed at baseline, 12 weeks and 6 months after initiation of the interventions.

Interventions:

1. IC: Participants visit the study site with health education, social activities, warm up, stretch, and low intensity resistance exercise for about 1 hour per week. If any medical problems or functional decline suspected during the visit, the case manager refers participants to their primary care physicians for further managements.
2. LEST: Participants receive 2 sessions of 30-minute lower extremity strength straining using isotonic strength training machines each week. The intensity is set at 60-80% of 1 repetition maximum (RM). Evaluation of the exercise protocol are repeated every 2 weeks for individualized adjustments

ELIGIBILITY:
Inclusion Criteria:

* Canadian Study of Health and Aging Clinical Frailty Scale (CSHA- CFS) Chinese In-Person Interview Version score is 3-6
* frailty index ≧ 1 (Cardiovascular Health Study Phenotypical Classification)。

Exclusion Criteria:

* age ≧ 80 years
* live in the nursing home.
* can not speak Chinese,Taiwanese.
* communication or hearing disorders affect daily activities.
* visual impairment or daily activities affect communication.
* another reason can not Communication or finish Canadian Study of Health and Aging Clinical Frailty Scale (CSHA- CFS) Chinese In-Person Version
* study of Health and Aging Clinical Frailty Scale (CSHA- CFS) Chinese In-Person Interview [9, 10]Version score is 0-2 and 7.
* communication or cognitive impairments affect daily activities(Exclusion 3-Item Recall score is <=1)
* can not stand to walk (available walkers) 5 meters, or unsteady gait when walking five meters, it looks fast fall
* there is serious risk of suicide (defined as: Suicide risk assessment score> = 6 points)
* alcoholism (defined as: the problem of alcoholism Chinese people self-administered screening questionnaire CAGE have two questions (including) above answer is "yes"
* long-term epilepsy, brain tumor, brain surgery, schizophrenia or bipolar disorder

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 98 (Actual)
Dates: Start 2011-03; Primary Completion 2011-03 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
leg extension power | changes in 12 weeks
  Leg extension power is to be measured at baseline, 12 weeks (after completion of intervention), and 6 months (after completion of the study). Specifically, following warm-up of three submaximal isotonic contractions, each subject was asked to extend his knee through a range of motions from -80 to -10 degrees of knee extension (0° extension being full knee extension without hyperextension) at an initial resistance equal to 25 percent of the subject's body weight. Knee range of motion was determined goniometrically. Following the successful completion of one full repetition, additional resistance of 1 kg, or a multiple thereof, was added. The repetition was repeated until the subject was no longer able to complete one full repetition. The number is the measured leg extension power

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Yu Chen, PHD, Study Chair — Department of Family MedicineNational Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan